CLINICAL TRIAL: NCT04738682
Title: Audit and Intervention of Diet Registration Method for Rehabilitation Patients at Hobro Hospital
Brief Title: Intervention of Diet Registration Method for Rehabilitation Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Movesca ApS (Unknown); Departmen for rehabilitation M3, Hobro Hospital (Unknown)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: AppHobro
Record Dates: First submitted 2021-01-25; First posted 2021-02-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Digital Clinical Diet Registrations Advantages; Patients in Rehabilitation
Keywords: dietary registration; methods for diet registration; comparison of electronic and paper registration

STUDY DESIGN:
Intervention Model Description: Modified crossover study model, containing two similar patient groups, exposed to identical diet registration methods, but in opposite sequence.
  Group 1: 3 days of digital dietary registration using mobile devices, followed by 3 days of conventional paper based dietary registration.
  Group 2: 3 days of conventional paper based dietary registration, followed by 3 days of digital dietary registration, using mobile devices.
  Each individual patient acts as his/her own control, with regards to the primary endpoint; precision. However patients are divided into two groups, in order to accommodate the study secondary endpoint; progression of nutritional condition, which is evaluated with regards to the registration method used. This requires two arms, where each arm experiences opposite registration method sequences
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Digital -> Conventional) (Active Comparator): Patients allocated to Group 1 (Digital -> Conventional) will undergo three days of digital dietary registration, using mobile devices, followed by three days of conventional dietary registration, using pen and paper.
  Interventions: Other: Digital dietary registration; Other: Conventional dietary registration
- Group 2 - (Conventional -> Digital) (Active Comparator): Patients allocated to Group 2 - (Conventional -> Digital) will undergo the exact opposite sequence, commencing with three days of conventional dietary registration, using pen and paper, followed by three days of digital dietary registration, using mobile devices.
  Interventions: Other: Digital dietary registration; Other: Conventional dietary registration

INTERVENTIONS:
Other: Digital dietary registration — The purpose of the intervention is to test whether digital dietary registration can yield more precise and consistent data, than conventional pen and paper based registration.
  Furthermore a subjective evaluation of the use of digital registration will be conducted by the staff upon completion of the intervention. The format will be individual interviews held by the investigators.
  Other Names: Dietary registration app supplied by Movesca ApS, used on cellphones present at the unit
Other: Conventional dietary registration — The conventional way of doing dietary registration. This is done by a paper form, with the dietary options listed. The form is then filled in and logged by staff working in the afternoon.
  Other Names: Paper form with all the possbible dietary options for each meal listed.

SUMMARY:
Study aims to investigate whether dietary registration can be performed with greater precision using digital registration units (mobile devices), rather than conventional paper based dietary registers.

Study intervention is based in the M3 rehabilitation unit, as part of Hobro hospital. The intervention will proceed until 6 full-day dietary registrations have been collected per patient (40 patients total), 3 for each registration method. The estimated time requirement is 30 days.

DETAILED DESCRIPTION:
Study aims to investigate whether dietary registration can be performed with greater precision using digital registration units (mobile devices), rather than conventional paper based dietary registers.

These mobile devices have been equipped with a dietary registration app, developed by the company Movesca ApS, specializing in digital healthcare solutions.

Nurses, and other relevant staff members at the M3 rehabilitation unit at Hobro hospital, will be testing this alternative registration method, as they engage in their day-to-day dietary registration for in-house patients. The data collection requires 6 full-day dietary registrations from each individual patient (40 patients in total). Of these 6 registrations, 3 will be gathered using mobile devices and 3 using conventional paper based registers.

The study primary endpoint is precision. The golden standard is dietary recall. The two methods will be assessed in accordance with their uniformity to the dietary recalls, which will be performed by the investigators following the meals.

As a preemptive measure, an internal retrospective audit was performed, with dietary registration as the objective. This audit was completed to retrieve baseline data on dietary registration, and determine whether the rehabilitation unit conforms to the regulations set by the region.

ELIGIBILITY:
Inclusion Criteria:

* The patient needs to be admitted to the rehabilitation unit at Hobro Hospital
* The patient need to give consent to be included.
* The patient needs to be admitted to the unit for at least 6 days
* The patient has to have 3 days of diet registration with both methods to be included in the data
* The patient need to be of legal age to give consent

Exclusion Criteria:

* The patient mustn be afflicted by any psychological illness, and must be of sound mind, so a normal conversation doesn't pose any problems.
* The patient mustn be sick with Covid-19, or other infectious diseases
* The patient mustn be terminal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Registered total kJ ingested compared to total kJ registered using golden standard | 4 weeks
  Does digital dietary registration yield greater precision than conventional paper based registration, in regards to total kJ?
Registered total protein ingested compared to total protein registered using golden standard | 4 weeks
  Does digital dietary registration yield greater precision than conventional paper based registration, in regards to protein intake?

SECONDARY OUTCOMES:
Is an adequate consumption of kJ (>75% of estimated kJ) achieved in fewer days with the digital dietary registration, than the conventional dietary registration | 4 weeks
  Do patients reach a stable nutritional state faster when exposed to digital dietary registration, compared to conventional paper based registration? Stable nutritional state is defined as consuming >75% of estimated kJ need per day. Tracked by comparing the registered consumed kJ of the day, with the estimated daily need
Is an adequate consumption of protein (>75% of estimated protein) achieved in fewer days with the digital dietary registration, than the conventional dietary registration | 4 weeks
  Do patients reach a stable nutritional state faster when exposed to digital dietary registration, compared to conventional paper based registration? Stable nutritional state is defined as consuming >75% of estimated protein need per day. Tracked by comparing the registered consumed protein of the day, with the estimated daily need

OTHER OUTCOMES:
Are the forms used for dietary registration filled out uniformly, by different personale | 4 weeks
  It will be examined whether or not the personal fills out the forms uniformly across all the included personale. It will be examined by comparing dietary registrations from different days, filled out by different personale.
Subjective experience of the staff regarding the intervention, examined by doing a semistructured interview with the personale. | 4 weeks
  Do staff consider digital dietary registration to be an improvement over conventional paper based registration? This will be explored by semistructured interview, held by the investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaj Nørlem, MSc, Principal Investigator — University of Copenhagen; Ted Rasmussen, MSc, Principal Investigator — University of Copenhagen
Locations (1):
- Department for rehabilitation medicine M3, Hobro, Denmark